CLINICAL TRIAL: NCT01403506
Title: Phase 3 Study of N-acetyl Cysteine as an Antioxidant and Glutathione Synthesis Inducer on Biomarkers of Delayed Renal Graft Function Including NGAL and IL-18
Brief Title: Study of the Effect of N-acetyl Cysteine on the Renal Graft Function Biomarkers (IL18, NGAL)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Jamshid Salamzadeh/Dr, Shaheed Beheshti Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 186
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-01

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: kidney transplantation; N-Acetyl Cysteine; living donor; delayed graft function
MeSH Terms: conditions — Delayed Graft Function | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Acetyl Cysteine (Active Comparator): N-Acetyl Cysteine: receive N-Acetyl Cysteine in addition to standard treatment
  Interventions: Drug: N-acetyl Cysteine
- standard treatment (No Intervention): This group is without N-Acetyl Cysteine : just receives standard treatment

INTERVENTIONS:
Drug: N-acetyl Cysteine — 600 mg N-acetyl Cysteine 6 hrs before renal transplantation, and 12 hrs and 18 hrs after renal transplantation.
  Other Names: Acetylcysteine; ACC 600
  Arms: N-Acetyl Cysteine

SUMMARY:
The purpose of this study is to investigate the effect of (NAC) N-Acetyl Cysteine on biomarkers of Delayed Graft Function (DGF), including Neutrophil Gelatinase Associated Lipocalin (NGAL) and Intereleukin 18 (IL18).

DETAILED DESCRIPTION:
Kidney transplantation is the best treatment for most patients with end stage renal failure, but limited numbers of suitable kidneys are available for transplantation. So preservation of graft is vital. This necessitates the studies and interventions to improve outcome of renal transplantation surgery.

Delayed Graft Function (DGF) or delay in performance of transplanted kidney means absence of acceptable function in the renal activity in postgrafting phase. DGF is a consequence of ischemic and reperfusion injuries (IRI), and oxygen free radicals have a main role in pathophysiology of DGF. In meta-analysis studies, it has been demonstrated that DGF has a correlation with long and short time graft survival. Despite great advances in the transplantation procedure, dysfunction prevalence has not decreased. Major causes of this problem are the lack of appropriate markers for early diagnosis of DGF and on the other hand lack of appropriate and effective interventions to controll DGF.

Studies have shown that N-Acetyl Cysteine (NAC) can induce GSH synthesis, scavenger of free radicals, and infusion of NAC had similar effects as glutathione.

This is a randomized clinical trial (RCT) on patients who have received kidney transplantation from living donors. Sixty transplanted patients will be randomized into 2 groups. The first group of patients will be treated with NAC 600mg 6 hr before transplantation and two doses of NAC 12 hours apart after transplantation in addition to standard treatment, and the second group will receive only standard antirejection treatment. For all patients entered the study, urinary concentrations of IL18 and NGAL will be measured in designated times. Risk factors of DGF will be compared in two groups and effectiveness of NAC in reducing DGF will be determined.

ELIGIBILITY:
Inclusion Criteria:

* patient receiving transplantation from living donors

Exclusion Criteria:

* having a neoplastic disease
* brain tumor
* having inflammatory diseases in their active phase (SLE)
* an acute infection, meningitis, sepsis
* Sickle Cell Disease
* Pregnancy
* Cardio-renal syndrome
* endogenous Cushing's syndrome
* chronic use of cimetidine
* a history of acute pancreatitis in recent months
* Multiple Sclerosis
* cardiac bypass in a recent month
* cirrhosis due to Hepatitis C
* having Alzheimer's disease
* having a untreated major depressive illness or schizophrenia
* Stroke in recent months
* Hyperoxaluria
* sensitivity to sulfonamides

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
renal function biomarkers (IL18, NGAL)difference between study and control group in 4 and 24 hr after transplantation | 4 and 24 hrs after renal graft

SECONDARY OUTCOMES:
dialysis | 60 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Jamshid Salamzadeh, PhD, Study Director — SBMU School of Pharmacy, Tehran, Iran
Locations (1):
- Department of Nephrology, Shahid Labbafinejad Medical Center and Urology and Nephrology Research Center, Shahid Beheshti University of Medical Sciences, Tehran, Tehran Province, Iran